CLINICAL TRIAL: NCT02111226
Title: DREAM-GLOBAL: Diagnosing hypeRtension - Engaging Action and Management in Getting LOwer Bp in Aboriginal and LMIC - A Research Proposal
Brief Title: Detecting and Treating High Blood Pressure in Aboriginal Population and Low and Middle Income Countries
Acronym: DREAM-GLOBAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Sheldon Tobe, Principal Investigator - Medical Doctor, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 182-2013
Record Dates: First submitted 2014-03-13; First posted 2014-04-11 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Hypertension; Cardiovascular Disease; Diabetes
Keywords: hypertension; cardiovascular disease; diabetes; chronic disease management
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Passive SMS Group (Active Comparator): Passive SMS messages focused on lifestyle adjustment
  Interventions: Other: SMS text messaging
- Active SMS Group (Experimental): Active SMS messages based on hypertension clinical practice guidelines including rational for taking antihypertensive medication and reminders to see the health care practioner if BP is above target.
  Interventions: Other: SMS text messaging

INTERVENTIONS:
Other: SMS text messaging — short message service

SUMMARY:
Heart disease and stroke are the number one killers world-wide. When someone has hypertension, the constantly elevated blood pressure damages their blood vessels and the organs that they supply blood to. This causes stroke, heart attack, heart failure, kidney failure and dementia. Finding and lowering high blood pressure to normal with lifestyle changes and if necessary medications, lowers the risk of these outcomes. Canada has high rates of blood pressure control compared to other countries in the world, due in large part to the successful dissemination of hypertension guidelines. However remote and disadvantaged communities have not been as successful and need additional measures to help achieve the same level of blood pressure control as the rest of the country. The DREAM-GLOBAL team has extensive experience working with Canada's Aboriginal Communities and a large community in Tanzania. The DREAM-GLOBAL project will integrate innovations in technology with the implementation of guidelines-based blood pressure control and through partnerships with experts in government and industry, overcome barriers to lowering blood pressure in Canada's Aboriginal Communities, and in a community in Tanzania. Tools will be developed and tested that will close the circle of care around people with hypertension by bringing measurement data to the medical record and health care provider and also sending useful medical feedback to the person with hypertension via secure data servers and routine SMS messaging on cell phones. The system will be tested for effectiveness of diagnosing and also for managing hypertension. To begin the process of preventing hypertension, the team will also explore with an Aboriginal community how to create policies to reduce the sodium content in their food. If proven effective, DREAM-GLOBAL can also become a platform for managing other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Hypertension
* BP > 140/90 mmHg or > 130/80 mmHg if patient has diabetes at the initial screening visit using an approved automated BP monitor.
* If on drug therapy, continuous drug therapy with the same dosing interval for 8 weeks prior to and throughout the screening period. May be drug naive.
* Written informed consent
* Hypertension for at least 12 weeks before screening and throughout the screening period (according to the patient or their medical practitioner)
* Must have a cell phone plan (in Canada) and be willing to maintain the plan during the study. For Tanzania, must have a cell phone under a locally available Tanzanian carrier.
* Must be willing to take occasional local calls from study team members
* One or more of BMI > 30 kg/m2, diabetes, smoking, over age 40, previous history of CAD including stroke and heart attack
* An identified health care provider in the community (ie. Family Physician/Nurse Practitioner in Canada or Community Nurse/Clinical officer in Tanzania)

Exclusion Criteria:

* Change in antihypertensive medication during the 8 weeks before enrolment
* No cell phone plan compatible with the study.
* Poorly controlled hypertension with BP > 180/110 mmHg
* No primary health care provider
* Active malignant disease (except non-melanoma skin cancer)
* Unable or unwilling to visit health care provider
* Unable to read the SMS messages (English in Canada and Kiswahili in Tanzania)
* Participation in a clinical trial or receipt of investigational compound or treatment in the 3 months prior to the initial screening visit.
* Planned elective surgery during the study period except for cataract surgery
* *For BP screening study, must not be on an antihypertensive in the last 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | one year
  The change in blood pressure (systolic and diastolic) from baseline to the final BP measurement period

SECONDARY OUTCOMES:
Blood Pressure | one year
  The proportion of patients achieving BP control during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon W Tobe, MD, MScCH (HPTE), FRCPC, FACP,, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto; Karen E Yeates, MD, FRCP(C), MPH, Principal Investigator — Queen's University; Norman RC Campbell, MD, FRCPC, Principal Investigator — University of Calgary; Peter Liu, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Barsky J, Hunter R, McAllister C, Yeates K, Campbell N, Liu P, Perkins N, Hua-Stewart D, Maar MA, Tobe SW. Analysis of the Implementation, User Perspectives, and Feedback From a Mobile Health Intervention for Individuals Living With Hypertension (DREAM-GLOBAL): Mixed Methods Study. JMIR Mhealth Uhealth. 2019 Dec 9;7(12):e12639. doi: 10.2196/12639. PMID 31815678
- [Derived] Maar MA, Beaudin V, Yeates K, Boesch L, Liu P, Madjedi K, Perkins N, Hua-Stewart D, Beaudin F, Wabano MJ, Tobe SW. Wise Practices for Cultural Safety in Electronic Health Research and Clinical Trials With Indigenous People: Secondary Analysis of a Randomized Clinical Trial. J Med Internet Res. 2019 Nov 4;21(11):e14203. doi: 10.2196/14203. PMID 31682574
- [Derived] Tobe SW, Yeates K, Campbell NRC, Maar MA, Perkins N, Liu PP, Sleeth J, McAllister C, Hua-Stewart D, Wells G, Bernick J. Diagnosing hypertension in Indigenous Canadians (DREAM-GLOBAL): A randomized controlled trial to compare the effectiveness of short message service messaging for management of hypertension: Main results. J Clin Hypertens (Greenwich). 2019 Jan;21(1):29-36. doi: 10.1111/jch.13434. Epub 2018 Nov 26. PMID 30474909
- [Derived] Yeates K, Campbell N, Maar MA, Perkins N, Liu P, Sleeth J, Smith C, McAllister C, Hua-Stewart D, Wells G, Tobe SW. The Effectiveness of Text Messaging for Detection and Management of Hypertension in Indigenous People in Canada: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Dec 19;6(12):e244. doi: 10.2196/resprot.7139. PMID 29258978
- [Derived] Maar MA, Yeates K, Perkins N, Boesch L, Hua-Stewart D, Liu P, Sleeth J, Tobe SW. A Framework for the Study of Complex mHealth Interventions in Diverse Cultural Settings. JMIR Mhealth Uhealth. 2017 Apr 20;5(4):e47. doi: 10.2196/mhealth.7044. PMID 28428165